CLINICAL TRIAL: NCT02202161
Title: A Randomized, Placebo Controlled, Repeat Dose, Double Blind (Sponsor Unblind) Study Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2330672 Administered With Metformin to Type 2 Diabetes Patients
Brief Title: A Study Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2330672 Administered With Metformin to Type 2 Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201351
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacokinetic; intestinal bile acid transporter inhibitor; metformin; sitagliptin; GSK2330672; pharmacodynamic
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((((3R,5R)-3-butyl-3-ethyl-7-(methyloxy)-1,1-dioxido-5-phenyl-2,3,4,5-tetrahydro-1,4-benzothiazepin-8-yl)methyl)amino)pentanedioic acid; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- GSK2330672 10 mg (Experimental): Subjects will receive metformin 850 mg BID for 13-15 days during the run in period followed by GSK2330672 10 mg BID for 14 days.
  Interventions: Drug: GSK2330672; Drug: Metformin
- GSK2330672 20 mg (Experimental): Subjects will receive metformin 850 mg BID for 13-15 days during the run in period followed by GSK2330672 20 mg BID for 14 days.
  Interventions: Drug: GSK2330672; Drug: Metformin
- GSK2330672 30 mg (Experimental): Subjects will receive metformin 850 mg BID for 13-15 days during the run in period followed by GSK2330672 30 mg BID for 14 days.
  Interventions: Drug: GSK2330672; Drug: Metformin
- GSK2330672 90 mg (Experimental): Subjects will receive metformin 850 mg BID for 13-15 days during the run in period followed by GSK2330672 90 mg BID for 14 days.
  Interventions: Drug: GSK2330672; Drug: Metformin
- GSK2330672-matched placebo (Placebo Comparator): Subjects will receive metformin 850 mg BID for 13-15 days during the run in period followed by matching placebo (of GSK2330672) BID for 14 days.
  Interventions: Drug: Placebo; Drug: Metformin
- Sitagliptin 50 mg (Active Comparator): Subjects will receive metformin 850 mg BID for 13-15 days during the run in period followed by Sitagliptin 50 mg BID for 14 days. In this study, sitagliptin 50 mg BID will be provided as open-label (unblinded) study treatment.
  Interventions: Drug: Sitagliptin; Drug: Metformin

INTERVENTIONS:
Drug: GSK2330672 — GSK2330672 will be available in 10 mg, 20 mg, 30 mg, and 90 mg oral solution to be administered BID for 14 days. Subjects are to drink contents of dosing bottle (45 ml) followed by 2 x 50 ml rinses of bottle and then an additional 95 ml water for a total volume of 240 ml consumed
  Arms: GSK2330672 10 mg; GSK2330672 20 mg; GSK2330672 30 mg; GSK2330672 90 mg
Drug: Placebo — Matching placebo will be available as oral solution to be administered for 14 days, BID. Subjects are to drink contents of dosing bottle (45 ml) followed by 2 x 50 ml rinses of bottle and then an additional 95 ml water for a total volume of 240 ml consumed
  Arms: GSK2330672-matched placebo
Drug: Sitagliptin — Sitagliptin will be available as film-coated tablets Tablet of 50 mg to be administered orally, BID, for 14 days
  Arms: Sitagliptin 50 mg
Drug: Metformin — Metformin will be available as 850 mg white to off-white, film-coated tablets; to be administered BID orally during run-in through Day 14

SUMMARY:
This study is being conducted to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of GSK2330672 compared to sitagliptin when administered with metformin for 14 days to subjects with type 2 diabetes mellitus (T2DM). Approximately 72 male and female subjects aged 30-64 years with T2DM and currently taking metformin will be recruited for this study. Eligible subjects will begin a run-in period of 13-15 days to stabilize on metformin 850 milligram (mg) twice a day (BID). Subjects will then be randomized to GSK2330672 10 mg, 20 mg, 30 mg, 90 mg, matching placebo or open-label sitagliptin 50 mg for 14 days BID. Subjects will return for a follow-up visit 7-10 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 30 and 64 years of age inclusive, at the time of signing the informed consent
* Subjects with a diagnosis of T2DM for at least 3 months prior to screening, taking metformin for at least 4 weeks prior to screening, taking a metformin daily dose of>= 1000 mg and having an Glycosolated haemoglobin A1c (HbA1c) value of 7-11% inclusive at screening. The investigator should make an effort to obtain documentation of medical history or prescription of metformin to substantiate the diagnosis of T2DM
* Fasting plasma glucose <280 milligram per deciliter (mg/dl) at screening. A subject with a fasting plasma glucose at Day 1 that is more than 100 mg/dl lower than the screening value must not be randomized
* All T2DM subjects must meet the label recommendations for metformin and sitagliptin, including: Adequate renal function, as evidenced by an estimated glomerular filtration rate >= 80 milliliter per minute (mL/min) using the modification of diet in renal disease (MDRD) equation or chronic kidney disease epidemiology collaboration (CKD-EPI) formula in the study procedures manual (SPM); No conditions which make hypoxia, dehydration, or sepsis likely; No cardiac disease (including no history of myocardial infarction, stroke, hospitalization for acute coronary syndrome, or heart failure)
* Body mass index (BMI) within the range 24 - 40 kilogram per meter square (kg/m^2) (inclusive)
* Other than T2DM, subjects should be in good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination that would introduce additional risk factors or interfere with study procedures or objectives, based on a medical evaluation including medical history, physical examination, vital signs, and laboratory tests
* A female subject is eligible to participate if she is of non-childbearing potential defined as: Pre-menopausal females with a documented tubal ligation, bilateral oophorectomy, or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; OR Postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 million international units (MlU)/mL and estradiol < 40 picogram (pg)/mL (<147 picomol per liter) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods as described by the Investigator/designee, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods as described by the Investigator/designee. This criterion must be followed from the time of the first dose of study medication until the follow-up visit
* Subjects must be willing to discontinue their usual dose of metformin and take the study dose of 850 mg immediate release formulation metformin BID for the 13-15 day run-in period and the 2-week treatment period
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* The use of approved non-metformin anti-diabetic agents within 3 months of the screening visit
* Hypoglycemia unawareness. T2DM subjects are excluded if, in the opinion of the investigator, they have significant hypoglycemia unawareness (for example, no symptoms of hypoglycemia when the blood glucose level is <70 mg/dl)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome). Subjects with a history of cholelithiasis, biliary colic, inflammatory gall bladder disease and/or cholestatic liver disease are excluded, unless this results in curative cholecystectomy 3 months or more before screening and with the approval of the GlaxoSmithKline (GSK) Medical Monitor
* History of chronic or acute pancreatitis. Approval from the GSK Medical Monitor must be obtained for subjects with a past history of pancreatitis more than 12 months from the start of the Treatment Period (subjects with a history of pancreatitis within 12 months prior to the start of the Treatment Period are excluded). NOTE: Subjects with a lipase value above the upper limit of normal (ULN) at screening are excluded. A single repeat assessment is allowed within 3 days of the original test
* History of Gastrointestinal (GI) disease (e.g., irritable bowel disease, chronic or current diarrhea, inflamed bowel, steatorrhoea/fat malabsorption, celiac disease, symptomatic lactose intolerance, small bowel resection). Subjects with gastroparesis requiring treatment are excluded. Subjects with history of prolapsed or bleeding haemorrhoids within 1 month of screening are excluded unless approved by the GSK Medical Monitor
* History of autonomic neuropathy
* History of epilepsy and/or use of anti-convulsants, including but not limited to phenobarbitone, phenytoin, carbamazepine, valproate
* History of serious, severe, or unstable physical or psychiatric illness including depression, suicidal thoughts, schizophrenia, bipolar disorder, or generalized anxiety disorder. In addition to elicited symptoms and signs, this should include specific questions relating to known psychiatric diagnoses and medications used
* History of significant cardiovascular disease not covered by the label recommendations for metformin, for example, ventricular tachyarrhythmias, peripheral arterial disease, and pulmonary embolism, within the previous 12 months
* Uncontrolled hypertension, as evidenced by systolic pressure >160 millimeters of mercury (mmHg) or diastolic pressure >90 mmHg on a single assessment. If systolic pressure >140 mmHg or diastolic pressure >90 mmHg, a single repeat is allowed within 1 hour. Subjects whose blood pressure is well-controlled by taking anti-hypertensive medications (e.g., beta blockers, angiotensin converting enzyme(ACE) inhibitors, angiotensin II receptor antagonists, calcium channel blockers, and thiazide diuretics) are permitted
* History of untreated pernicious anemia or who have laboratory parameters suggestive of subclinical megaloblastic anemia (e.g., increased mean corpuscular volume [MCV] with low red blood cells [RBC] count and/or haemoglobin [Hb] level).
* Thyroid disease: Uncorrected Thyroid Dysfunction as Fasting plasma thyroid stimulating hormone (TSH) outside of the normal range, as determined at the screening visit. Subjects on stable thyroid replacement therapy and with TSH in the normal range are eligible if approved by the GSK Medical Monitor. Unevaluated thyroid nodule or goiter at screening
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy (including other Dipeptidyl Peptidase-IV [DPP-IV] inhibitors) that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Current or relevant previous significant medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that, in the opinion of the investigator, presents undue risk from the study medication or procedures
* Alanine aminotransferase (ALT)>2xULN and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Fasting triglycerides >= 400 mg/dl for subjects without a history of pancreatitis or >250 mg/dl for subjects with a history of pancreatitis. Approval from the GSK Medical Monitor must be obtained for subjects with a past history of pancreatitis more than 12 months from the start of the treatment period (subjects with a history of pancreatitis within 12 months prior to the start of the treatment period are excluded). Subjects taking statins, ezetimibe, or Vytorin are permitted in the study. Subjects taking other lipid therapies, including but not limited to niacin, bile acid sequestrants and/or fibrates are not eligible
* C-peptide of <0.8 nanogram (ng)/mL at screening
* Urine albumin-to-creatinine ratio >0.3 mg albumin/mg creatinine
* Positive fecal occult blood test at screening or during the run-in period
* Significant ECG abnormalities, defined as follows: Heart Rate (resting) was <50 and >100 beats per minute (bpm); PR Interval between <120 and >220 millisecond (msec); QRS duration between <70 and >120 msec
* Based on averaged QTcF of triplicate ECGs obtained at least 1 minute apart within approximately 15 minutes: QT duration corrected for heart rate by Fridericia's formula (QTcF) >= 450 msec; OR QTcF >= 480 msec in subjects with right Bundle Branch Block (subjects with left bundle branch block are excluded)
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody
* A positive urine drug screen or alcohol breath test at screening or during the run-in or treatment periods
* A subject with a positive urine cotinine test result will be excluded from the study unless in the judgment of the investigator the subject will be able to abstain from using tobacco for the duration of the in-clinic treatment period of the study
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Subjects who have participated in a previous study with GSK2330672 are excluded
* Because of the potential impact on bile acid synthesis and secretion in the liver, use of rifampicin and/or other pregnane X receptor (PXR) inducers, including but not limited to St. John's Wort, is cause for subject exclusion

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 201351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 27 August 2014 to 30 January 2015. After interim analysis of safety, tolerability, pharmacodynamic and/or pharmacokinetic (PK) data, GSK2330672 10 and 20 milligram (mg) doses were dropped and GSK2330672 60 mg was added.
Pre-assignment Details: A total of 187 participants were screened, of these, 112 were screen failures and 75 entered the run-in period. Five participants were withdrawn prior to taking a metformin dose in the 14 days of run-in period. A total of 64 participants were randomized to receive investigational product, as 6 participants were withdrawn prior to randomization.
Groups:
- Placebo: Participants were randomized to receive matching placebo solution of GSK2330672 orally twice daily (BID) for 14 days. Participants drank the contents of dosing bottle (45 milliliters [mL]) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The matching placebo solution of GSK2330672, was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued to receive metformin 850 mg BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
- GSK2330672 10 mg BID: Participants were randomized to receive solution of GSK2330672 10 mg orally BID for 14 days. Participants drank the contents of dosing bottle (45 mL) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The solution of GSK2330672 (2 mg/mL), was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued to receive metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
- GSK2330672 20 mg BID: Participants were randomized to receive solution of GSK2330672 20 mg orally BID for 14 days. Participants drank the contents of dosing bottle (45 mL) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The solution of GSK2330672 (2 mg/mL), was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued received metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
- GSK2330672 30 mg BID: Participants were randomized to receive solution of GSK2330672 30 mg orally BID for 14 days. Participants drank the contents of dosing bottle (45 mL) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The solution of GSK2330672 (2 mg/mL), was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued to receive metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
- GSK2330672 60 mg BID: Participants were randomized to receive solution of GSK2330672 60 mg orally BID for 14 days. Participants drank the contents of dosing bottle (45 mL) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The solution of GSK2330672 (2 mg/mL), was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued to receive metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
- GSK2330672 90 mg BID: Participants were randomized to receive solution of GSK2330672 90 mg orally BID for 14 days. Participants drank the contents of dosing bottle (45 mL) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The solution of GSK2330672 (2 mg/mL), was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued to receive metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
- Sitagliptin 50 mg BID: Participants were randomized to receive sitagliptin 50 mg tablet orally BID for 14 days. Participants continued to receive metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the both whole tablets of sitagliptin and metfornin with 240 mL of water each and were instructed to avoid chewing or crushing.
- Run-in Only: Participants were received open label metformin 850 mg tablet BID during run-in period, but were withdrawn prior to randomization. Participants swallowed the whole tablet with 240 mL of water and were instructed to avoid chewing or crushing.
Period: Overall Study
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID | Run-in Only
Started | 13 | 5 | 5 | 9 | 9 | 10 | 13 | 6
Completed | 12 | 4 | 5 | 9 | 8 | 9 | 13 | 0
Not Completed | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 6
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Did not meet continuation criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were randomized to receive matching placebo solution of GSK2330672 orally BID for 14 days. Participants drank the contents of dosing bottle (45 mL) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The matching placebo solution of GSK2330672, was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued to receive metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID | Run-in Only | Total
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13 | 6 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (6.97) | 54.0 (4.30) | 56.2 (8.50) | 57.1 (5.86) | 55.0 (4.27) | 54.8 (7.47) | 53.7 (6.79) | 55.5 (3.51) | 54.5 (6.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 2 | 6 | 4 | 5 | 3 | 31
  Male | 9 | 2 | 1 | 7 | 3 | 6 | 8 | 3 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
  Black or African American | 3 | 1 | 0 | 1 | 3 | 0 | 3 | 1 | 12
  White | 10 | 4 | 4 | 8 | 4 | 9 | 10 | 5 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Derived Plasma Glucose Parameter Over a 24-hour Period-fasting and Weighted Mean Glucose Area Under Curve (AUC[0-24 Hour])
Description: The change from Baseline was calculated by subtracting the Baseline values from the individual post-Baseline values. Baseline was defined as pre-dose Day -1 value. It was assessed on Baseline, Day 7 and 14. Data for fasting and weighted mean (WM) AUC(0-24 hour) glucose is provided. Statistics for least square mean is provided and participants withdrawing early were excluded. Results were based on an analysis of covariance (ANCOVA) model: change from Baseline = Baseline + treatment.
Time Frame: Baseline (Day -1) and Day 14 (Fasting Pre-dose [within 15 minutes of dose], 30 minutes, 1, 1.5, 2, 4 [pre-lunch], 5.5, 10 [pre-dinner], 11.5, 14 [bed time] and 24 hours) and Day 7 (30 minutes, 2, 4 [pre-lunch], 5.5, 10 [pre-dinner], 11.5, and 24 hours)
Population: Safety population was used which was defined as all participants enrolled into the study who received at least one dose of study drug (including GSK2330672, GSK2330672-matched placebo, sitagliptin and metformin). Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Mg/deciliter
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Mg/deciliter
  Fasting, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  Fasting, Day 7 | -6.58 (16.357) | -8.25 (6.500) | -1.40 (23.050) | -38.56 (24.744) | -34.38 (19.398) | -24.78 (13.414) | -24.54 (33.955)
  Fasting, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  Fasting, Day 14 | -10.00 (19.207) | -22.75 (11.354) | -16.20 (28.709) | -48.67 (32.650) | -36.13 (23.117) | -40.22 (19.156) | -38.38 (16.439)
  WM AUC(0-24 hour), Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  WM AUC(0-24 hour), Day 7 | 3.91 (20.668) | -12.14 (11.828) | -7.01 (17.262) | -25.33 (25.819) | -21.47 (18.419) | -14.84 (18.569) | -26.63 (23.610)
  WM AUC(0-24 hour), Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  WM AUC(0-24 hour), Day 14 | -9.94 (18.458) | -22.44 (15.928) | -17.80 (16.990) | -37.48 (32.909) | -32.22 (22.948) | -45.54 (21.010) | -35.85 (20.233)
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — An analysis of covariance (ANCOVA) model with a fixed effect term for treatment was fitted with the post-Baseline pharmacodynamic parameter value minus Baseline (Day -1 parameter value) as the dependent variable and Baseline as a covariate; Mean Difference (Net) = -1.17, 95% CI 2-sided [-25.61 to 23.27] — Comparison for fasting, Day 7
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 13.22, 95% CI 2-sided [-9.84 to 36.27] — Comparison for fasting, Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -21.77, 95% CI 2-sided [-41.43 to -2.10] — Comparison for fasting, Day 7
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -23.10, 95% CI 2-sided [-42.63 to -3.57] — Comparison for fasting, Day 7
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -11.79, 95% CI 2-sided [-30.85 to 7.28] — Comparison for fasting, Day 7
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -10.04, 95% CI 2-sided [-27.66 to 7.57] — Comparison for fasting, Day 7
Statistical Analysis 7: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -15.14, 95% CI 2-sided [-37.72 to 7.43] — Comparison for WM AUC(0-24 hour), Day 7
Statistical Analysis 8: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.10, 95% CI 2-sided [-23.66 to 19.45] — Comparison for WM AUC(0-24 hour), Day 7
Statistical Analysis 9: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -20.66, 95% CI 2-sided [-38.75 to -2.57] — Comparison for WM AUC(0-24 hour), Day 7
Statistical Analysis 10: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -21.70, 95% CI 2-sided [-39.70 to -3.71] — Comparison for WM AUC(0-24 hour), Day 7
Statistical Analysis 11: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -10.62, 95% CI 2-sided [-28.62 to 7.38] — Comparison for WM AUC(0-24 hour), Day 7
Statistical Analysis 12: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -26.03, 95% CI 2-sided [-41.94 to -10.12] — Comparison for WM AUC(0-24 hour), Day 7
Statistical Analysis 13: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -12.10, 95% CI 2-sided [-33.56 to 9.36] — Comparison for fasting, Day 14
Statistical Analysis 14: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.33, 95% CI 2-sided [-15.91 to 24.57] — Comparison for fasting, Day 14
Statistical Analysis 15: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -25.29, 95% CI 2-sided [-42.56 to -8.02] — Comparison for fasting, Day 14
Statistical Analysis 16: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -19.97, 95% CI 2-sided [-37.12 to -2.82] — Comparison for fasting, Day 14
Statistical Analysis 17: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -21.82, 95% CI 2-sided [-38.56 to -5.08] — Comparison for fasting, Day 14
Statistical Analysis 18: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -18.01, 95% CI 2-sided [-33.48 to -2.55] — Comparison for fasting, Day 14
Statistical Analysis 19: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -11.20, 95% CI 2-sided [-33.21 to 10.81] — Comparison for WM AUC(0-24 hour), Day 14
Statistical Analysis 20: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.80, 95% CI 2-sided [-16.22 to 25.81] — Comparison for WM AUC(0-24 hour), Day 14
Statistical Analysis 21: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -15.23, 95% CI 2-sided [-32.86 to 2.41] — Comparison for WM AUC(0-24 hour), Day 14
Statistical Analysis 22: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -17.01, 95% CI 2-sided [-34.56 to 0.53] — Comparison for WM AUC(0-24 hour), Day 14
Statistical Analysis 23: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -23.94, 95% CI 2-sided [-41.49 to -6.39] — Comparison for WM AUC(0-24 hour), Day 14
Statistical Analysis 24: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -19.45, 95% CI 2-sided [-34.96 to -3.93] — Comparison for WM AUC(0-24 hour), Day 14

2. Primary Outcome: Number of Participants With Incidence and Nature of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition and alanine aminotransferase (ALT) >= 3× upper limit of normal (ULN) and total bilirubin >=2 × ULN (>35% direct) or ALT >=3 × ULN and international normalized ratio >1.5.
Time Frame: Up to 14 days (treatment period)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Participants
  Any AE | 9 | 4 | 5 | 5 | 8 | 8 | 8
  Any SAE | 0 | 1 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Hematology With Potential Clinical Concern (PCI)
Description: Hematology parameters included platelet, red blood cell (RBC) count, mean corpuscular volume (MCV), neutrophils, white blood cell (WBC) count (absolute), mean corpuscular hemoglobin (MCH), lymphocytes, mean corpuscular hemoglobin concentration (MCHC), monocytes, hemoglobin, eosinophils, hematocrit and basophils. It was assessed on Baseline (pre-dose Day -1), Day 7 and 15. Data for parameters with above and below the PCI is provided.
Time Frame: Up to Day 15
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry With PCI
Description: Clinical chemistry parameters included blood urea nitrogen (BUN), potassium, aspartate aminotransferase (AST), total bilirubin, direct bilirubin, creatinine, chloride, alanine aminotransferase (ALT), uric acid, fasting glucose, total carbon dioxide, gamma glutamyltransferase (GGT), albumin, sodium, calcium, alkaline phosphatase (ALP), total protein, total carbon dioxide and triglycerides. It was assessed on Baseline (pre-dose Day -1), Day 7 and 15. Data for parameters with above and below the PCI is provided. The normal range (NR) and PCI definition for abnormal parameters are: ALT (NR: 0-44, 0-32, 2-33; PCI: >=2×upper limit of normal [ULN]); AST (NR: 0-40; PCI: >=2× ULN) and total bilirubin (NR: 0.00-20.52; PCI: >=1.5× ULN).
Time Frame: Up to Day 15
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Participants
  ALT, high | 1 | 0 | 2 | 2 | 2 | 1 | 1
  AST, high | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Total Bilirubin, hgh | 0 | 0 | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Urinalysis Data
Description: Urinalysis included urine occult blood: trace to 3+, glucose: negative to 3+, protein: negative to 2+ and ketones: trace to negative by dipstick and microscopic examination included cast, cellular cast, granular cast, hyaline cast (none seen to 1) and RBC: 0-2, 3-10, 11-30, >30, WBC: none seen, 0-5, 1, 2, 4, <5, 6-10, 11-30, 19, >30). The plus sign increases with a higher level of occult blood, glucose, ketones, proteins, RBC, WBC in the urine: 1+: slightly positive, 2+: positive, 3+: high positive. Participants were categorized as none seen or 1 based on the absence or presence, respectively, of cast, cellular cast, granular cast and hyaline cast. Higher value indicates higher abnormality.
Time Frame: Baseline (pre-dose Day -1), Day 7 and 15
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Participants
  Urine Occult Blood, Day -1, Trace | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Urine Occult Blood, Day -1, small | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Occult Blood, Day-1, 3+ | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Urine Occult Blood, Day 7, Trace | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Urine Occult Blood, Day 7, Trace intact | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Occult Blood, Day 7, small | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Occult Blood, Day 7, 1+ | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Occult Blood, Day 15, Trace | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Occult Blood, Day 15, small | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Occult Blood, Day 15, 2+ | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Microscopy-Casts, Day 7, none seen | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-Cellular Casts, Day -1, none seen | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Urine Microscopy-Cellular Casts, Day 7, none seen | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Urine Microscopy-Cellular Casts, Day 15, none seen | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Urine Microscopy-Granular Casts, Day -1, none seen | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Urine Microscopy-Granular Casts, Day 7, none seen | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Urine Microscopy-Granular Casts, Day 15, none seen | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Urine Glucose, Day -1, Trace | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Urine Glucose, Day -1, 1+ | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Urine Glucose, Day -1, 2+ | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Glucose, Day -1, 3+ | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Urine Glucose, Day 7, Trace | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Urine Glucose, Day 7, 1+ | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Urine Microscopy-Hyaline Casts, Day -1, none seen | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Urine Microscopy-Hyaline Casts, Day 7, None seen | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Urine Microscopy-Hyaline Casts, Day 7, 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Microscopy-Hyaline Casts, Day 15, none seen | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Urine Ketones, Day 7, Trace | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urine Protein, Day -1, 1+ | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urine Protein, Day 7, 2+ | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urine Protein, Day 15, Trace | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Urine Protein, Day 15, 1+ | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urine Microscopy-RBC, Day -1, none seen | 2 | 0 | 0 | 1 | 0 | 0 | 1
  Urine Microscopy-RBC, Day -1, 0-2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-RBC, Day -1, 3-10 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Urine Microscopy-RBC, Day -1, 11-30 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Urine Microscopy-RBC, Day 7, none seen | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Urine Microscopy-RBC, Day 7, 0-2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Urine Microscopy-RBC, Day 15, none seen | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Urine Microscopy-RBC, Day 7, 3-10 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day -1, none seen | 2 | 2 | 0 | 1 | 0 | 0 | 1
  Urine Microscopy-WBC, Day -1, 0-5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Microscopy-WBC, Day -1, 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Microscopy-WBC, Day -1, 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day -1, 6-10 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urine Microscopy-WBC, Day -1, 11-30 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day -1, >30 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day 7, 0-5 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Urine Microscopy-WBC, Day 7, 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Urine Microscopy-WBC, Day 7, <5 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day 7, 11-30 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Urine Microscopy-WBC, Day 7, 19 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day 7, >30 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day 15, 0-5 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Urine Microscopy-WBC, Day 15, 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day 15, 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Microscopy-WBC, Day 15, 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Microscopy-WBC, Day 15, 11-30 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urine Microscopy-WBC, Day 15, >30 | 0 | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Summary of Urinalysis Data-mean Specific Gravity
Description: Data for mean specific gravity is provided. Specific gravity is a measure of the amount of material dissolved in the urine. Specific gravity is the ratio of the density (mass of a unit volume) of a substance to the density (mass of the same unit volume) of a reference substance. Normal urine has a specific gravity between 1.010 and 1.020.
Time Frame: Baseline (pre-dose Day -1), Day 7 and 15
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Ratio
  Day -1 | 1.0193 (0.00694) | 1.0182 (0.00581) | 1.0128 (0.00421) | 1.0190 (0.00618) | 1.0172 (0.00610) | 1.0189 (0.00780) | 1.0148 (0.00706)
  Day 7: number analyzed (Participants) | 12 | 5 | 5 | 9 | 8 | 10 | 13
  Day 7 | 1.0196 (0.00753) | 1.0208 (0.00904) | 1.0184 (0.00896) | 1.0191 (0.00739) | 1.0194 (0.00726) | 1.0208 (0.00859) | 1.0160 (0.00790)
  Day 15: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 9 | 13
  Day 15 | 1.0188 (0.00403) | 1.0193 (0.00435) | 1.0158 (0.00259) | 1.0132 (0.00471) | 1.0121 (0.00348) | 1.0160 (0.00787) | 1.0140 (0.00815)

7. Primary Outcome: Summary of Urinalysis Data-mean pH
Description: Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Baseline (pre-dose Day -1), Day 7 and 15
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Unit on a scale
  Day -1 | 5.73 (0.388) | 6.00 (0.000) | 6.10 (0.224) | 6.11 (0.220) | 5.83 (0.354) | 5.95 (0.438) | 5.85 (0.516)
  Day 7: number analyzed (Participants) | 12 | 5 | 5 | 9 | 9 | 10 | 13
  Day 7 | 5.83 (0.389) | 5.90 (0.224) | 6.00 (0.000) | 5.89 (0.220) | 5.61 (0.486) | 5.95 (0.284) | 5.69 (0.435)
  Day 15: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 9 | 13
  Day 15 | 5.88 (0.377) | 5.88 (0.250) | 6.00 (0.000) | 6.00 (0.000) | 5.72 (0.565) | 6.06 (0.167) | 5.88 (0.416)

8. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings Any Time Post-Baseline
Description: Single 12-lead ECGs was obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. It was assessed on Baseline (pre-dose Day -1), Day 7 and 15. Participants with normal, abnormal not clinically significant and abnormal clinically significant ECG is presented.
Time Frame: Up to Day 15
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Participants
  Normal | 9 | 4 | 4 | 8 | 6 | 6 | 9
  Abnormal not clinically significant | 4 | 0 | 1 | 1 | 3 | 4 | 4
  Abnormal clinically significant | 0 | 1 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Change From Baseline in Vital Signs Assessments-temperature
Description: The change from Baseline was calculated by subtracting the Baseline values from the individual post-Baseline values. Baseline was defined as pre-dose Day -1 value.
Time Frame: Baseline (pre-dose Day -1) and, Day 7, 15
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Degree Celsius
  Day 7: number analyzed (Participants) | 12 | 5 | 5 | 9 | 9 | 10 | 13
  Day 7 | -0.133 (0.2570) | -0.280 (0.4764) | 0.040 (0.4393) | 0.033 (0.3937) | 0.033 (0.2062) | 0.010 (0.4458) | 0.015 (0.4451)
  Day 15: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 9 | 13
  Day 15 | -0.208 (0.3370) | 0.025 (0.1708) | -0.040 (0.2966) | -0.111 (0.5622) | 0.056 (0.2744) | -0.178 (0.5995) | 0.062 (0.3404)

10. Primary Outcome: Change From Baseline in Vital Signs Assessments-systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: as for outcome 9
Time Frame: Baseline (pre-dose Day -1) and Day 7, 15
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Millimeters of mercury
  DBP, Day 7: number analyzed (Participants) | 12 | 5 | 5 | 9 | 9 | 10 | 13
  DBP, Day 7 | -0.083 (6.8152) | -1.600 (8.5323) | -6.600 (1.9494) | -1.556 (10.7948) | -4.111 (4.9861) | -2.700 (6.7007) | -2.462 (7.6770)
  DBP, Day 15: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 9 | 13
  DBP, Day 15 | 0.750 (6.1070) | -2.750 (4.5735) | 1.800 (5.8481) | -1.333 (9.1104) | -1.667 (3.9370) | -2.667 (6.3048) | -0.769 (5.0852)
  SBP, Day 7: number analyzed (Participants) | 12 | 5 | 5 | 9 | 9 | 10 | 13
  SBP, Day 7 | 2.250 (8.4544) | -4.000 (10.2225) | -15.600 (6.1482) | 2.222 (17.6973) | 1.222 (9.1211) | -4.300 (10.9245) | -5.462 (10.3571)
  SBP, Day 15: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 9 | 13
  SBP, Day 15 | 2.167 (8.5049) | -4.500 (10.4722) | 0.600 (11.8870) | -5.111 (11.9105) | -1.000 (9.3541) | -2.111 (9.5321) | -4.385 (9.2334)

11. Primary Outcome: Change From Baseline in Vital Signs Assessments-heart Rate
Description: as for outcome 9
Time Frame: Baseline (pre-dose Day -1) and Day 7, 15
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Beats per minute
  Day 7: number analyzed (Participants) | 12 | 5 | 5 | 9 | 9 | 10 | 13
  Day 7 | -0.500 (8.1296) | 9.200 (8.2280) | 4.400 (7.4027) | 0.556 (5.2941) | 4.667 (4.0620) | 1.400 (7.0269) | -0.769 (6.2471)
  Day 15: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 9 | 13
  Day 15 | 0.083 (3.1176) | 0.250 (6.3443) | 9.200 (3.1937) | -0.444 (8.2932) | 4.889 (7.4237) | 0.000 (8.8034) | 1.846 (9.1364)

12. Primary Outcome: Number of Bowel Movements (Stool Frequency) as Rated Using the Bristol Stool Form Scale (BSFS) Across Days 1 to 14
Description: The site staff classified participant's stools and record the date and time of occurrence after any bowel movement that occurs while participants were in residence in the clinic. BSFS is scale between type 1-7, it measured the shape of the stool, type 1: separate hard lumps, like nuts; type 2: sausage shaped but lumpy; type 3: like a sausage or snake but with cracks on its surface; type 4: like a sausage or snake, smooth and soft; type 5: soft blobs with clear cut edges; type 6: fluffy pieces with ragged edges, a mushy stool and type 7: watery, no solid pieces. Participants were discharged after they have had at least one bowel movement after the Day 14 dosing and after the investigator/designee had reviewed the Day 15 end of study questions.
Time Frame: Up to Day 15 (administered after every in-house bowel movement)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Count of bowel movements
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID | Run-in Only
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13 | 0
Count of bowel movements | 15.2 (9.29) | 28.2 (17.47) | 38.4 (10.74) | 35.0 (18.49) | 37.3 (30.72) | 35.9 (21.67) | 15.0 (10.96) |

13. Primary Outcome: Number of Events With the Rating on Quality of Stools as Rated Using the BSFS Across Days 1 to 14
Description: as for outcome 12
Time Frame: Up to Day 15 (administered after every in-house bowel movement)
Population: Safety population. Only those participants available at the specified time points were analyzed. For each BSFS scale rating the "Number of Participants Analyzed" represents the number of participants reporting that rating not the number evaluated.
Measure: Number; unit: Events
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Events
  BSFS scale rating, 1 event : Events: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 1 | 2
  BSFS scale rating, 1 event : Events | 2 |  |  | 1 |  | 1 | 2
  BSFS scale rating, 2 events : Events: number analyzed (Participants) | 2 | 0 | 2 | 1 | 0 | 0 | 7
  BSFS scale rating, 2 events : Events | 6 |  | 2 | 1 |  |  | 10
  BSFS scale rating, 3 events : Events: number analyzed (Participants) | 5 | 0 | 2 | 1 | 3 | 5 | 10
  BSFS scale rating, 3 events : Events | 28 |  | 4 | 1 | 6 | 5 | 36
  BSFS scale rating, 4 events : Events: number analyzed (Participants) | 11 | 2 | 5 | 6 | 6 | 8 | 9
  BSFS scale rating, 4 events : Events | 56 | 7 | 18 | 19 | 21 | 24 | 41
  BSFS scale rating, 5 events : Events: number analyzed (Participants) | 8 | 2 | 4 | 7 | 3 | 9 | 9
  BSFS scale rating, 5 events : Events | 30 | 2 | 8 | 26 | 9 | 30 | 26
  BSFS scale rating, 6 events : Events: number analyzed (Participants) | 9 | 5 | 5 | 9 | 8 | 10 | 9
  BSFS scale rating, 6 events : Events | 59 | 81 | 113 | 181 | 250 | 201 | 70
  BSFS scale rating, 7 events : Events: number analyzed (Participants) | 7 | 4 | 5 | 8 | 7 | 8 | 3
  BSFS scale rating, 7 events : Events | 16 | 51 | 47 | 86 | 50 | 98 | 10

14. Primary Outcome: Number of Participants With Gastrointestinal Tolerability Assessments as Rated Using the Gastrointestinal Symptom Rating Scale (GSRS; With Worsening Symptoms >=2 Levels)
Description: GSRS is a rating scale consisting of 15 items. Each item was scored from 1: no discomfort at all, 2: minor discomfort, 3: mild discomfort, 4: moderate discomfort, 5: moderately severe discomfort, 6: severe discomfort, 7: very severe discomfort. The overall GSRS score is the mean of these 15 items, varying from 1 to 7; a score of 1 indicates that no symptoms are present, and a score of 7 indicates the worst possible degree of all symptoms. A higher score relative to Baseline indicates worsening of severity. There were 5 defined syndrome scores and 1 overall score that was derived by computing the mean of the scores for specific subsets of questions as indicated below: abdominal pain (1, 4, 5); reflux syndrome (2, 3); diarrhea syndrome (11, 12, 14); indigestion syndrome (6, 7, 8, 9); constipation syndrome (10, 13, 15) and overall GSRS (1-15). The data is presented for participants with worsening of symptoms in >=2 levels.
Time Frame: Day 7 and 14
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Participants
  Pain/discomfort in upper abdomen, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Pain/discomfort in upper abdomen, Day 7 | 0 | 0 | 2 | 2 | 0 | 0 | 0
  Heartburn, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Heartburn, Day 7 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Acid reflux, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Acid reflux, Day 7 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Hunger pains, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Hunger pains, Day 7 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  Nausea, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Nausea, Day 7 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Rumbling, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Rumbling, Day 7 | 1 | 0 | 2 | 0 | 1 | 2 | 0
  Bloated, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Bloated, Day 7 | 2 | 0 | 1 | 1 | 0 | 3 | 0
  Burping, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Burping, Day 7 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  Passing gas or flatus, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Passing gas or flatus, Day 7 | 1 | 1 | 1 | 1 | 0 | 2 | 0
  Constipation, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Constipation, Day 7 | 1 | 0 | 3 | 4 | 3 | 0 | 0
  Diarrhea, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Diarrhea, Day 7 | 0 | 0 | 2 | 3 | 4 | 4 | 0
  Loose stools, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Loose stools, Day 7 | 1 | 0 | 3 | 4 | 3 | 3 | 0
  Hard stools, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Hard stools, Day 7 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Urgent need to have bowel movement, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Urgent need to have bowel movement, Day 7 | 1 | 0 | 2 | 1 | 2 | 2 | 0
  Sensatn not complete empty bowels, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Sensatn not complete empty bowels, Day 7 | 0 | 0 | 2 | 2 | 3 | 2 | 0
  Abdominal pain, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Abdominal pain, Day 7 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Reflux syndrome, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Reflux syndrome, Day 7 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Indigestion syndrome, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Indigestion syndrome, Day 7 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  Constipation syndrome, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Constipation syndrome, Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea syndrome, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Diarrhea syndrome, Day 7 | 0 | 0 | 2 | 3 | 2 | 2 | 0
  Overall GSRS, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 9 | 10 | 13
  Overall GSRS, Day 7 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Pain/discomfort in upper abdomen, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Pain/discomfort in upper abdomen, Day 14 | 1 | 1 | 2 | 1 | 1 | 1 | 1
  Heartburn, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 10
  Heartburn, Day 14 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Acid reflux, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Acid reflux, Day 14 | 1 | 1 | 1 | 0 | 0 | 1 | 0
  Hunger pains, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Hunger pains, Day 14 | 0 | 0 | 2 | 2 | 0 | 2 | 0
  Nausea, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Nausea, Day 14 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Rumbling, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Rumbling, Day 14 | 1 | 1 | 2 | 1 | 0 | 2 | 0
  Bloated, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Bloated, Day 14 | 2 | 1 | 2 | 1 | 0 | 3 | 00
  Burping, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Burping, Day 14 | 1 | 1 | 1 | 0 | 0 | 2 | 0
  Passing gas or flatus, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Passing gas or flatus, Day 14 | 0 | 1 | 2 | 2 | 0 | 2 | 0
  Constipation, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Constipation, Day 14 | 0 | 1 | 1 | 0 | 0 | 2 | 0
  Diarrhea, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Diarrhea, Day 14 | 1 | 0 | 4 | 3 | 2 | 5 | 0
  Loose stools, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Loose stools, Day 14 | 1 | 1 | 3 | 2 | 3 | 3 | 0
  Hard stools, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Hard stools, Day 14 | 0 | 0 | 2 | 0 | 0 | 1 | 0
  Urgent need to have bowel movement, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Urgent need to have bowel movement, Day 14 | 1 | 1 | 4 | 2 | 3 | 3 | 0
  Sensation not complete empty bowels, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Sensation not complete empty bowels, Day 14 | 0 | 0 | 3 | 2 | 3 | 2 | 0
  Abdominal pain, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Abdominal pain, Day 14 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Reflux syndrome, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Reflux syndrome, Day 14 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  Indigestion syndrome, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Indigestion syndrome, Day 14 | 0 | 1 | 1 | 1 | 0 | 2 | 0
  Constipation syndrome, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Constipation syndrome, Day 14 | 0 | 0 | 2 | 0 | 0 | 2 | 0
  Diarrhea syndrome, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Diarrhea syndrome, Day 14 | 0 | 0 | 3 | 2 | 1 | 3 | 0
  Overall GSRS, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 10 | 13
  Overall GSRS, Day 14 | 0 | 0 | 1 | 1 | 0 | 2 | 0

15. Primary Outcome: Number of Participants With Fecal Occult Blood Monitoring for Symptomatic or Visible Gastrointestinal Bleeding or Asymptomatic Occult Bleeding
Description: Testing cards were provided to participants for assessments. Participants with abnormal not clinically significant and abnormal clinically significant is presented. The Day -1 sample was obtained any time starting Day -2 and prior to GSK2330672 dosing on Day 1. The Day 14 sample was collected any time after dosing on Day 14 and prior to discharge on Day 15.
Time Frame: Up to Day 15
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID | Run-in Only
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13 | 6
Participants
  Abnormal not clinically significant | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  Abnormal clinically significant | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

16. Secondary Outcome: PK Parameters for Metformin Steady State PK Parameters When Co-dosed With GSK2330672, Sitagliptin or Placebo-maximum Observed Concentration (Cmax)
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. Statistics for geometric least square mean provided.
Time Frame: Fasting pre-dose (within 15 minutes of dose), 30 minutes, 1, 1.5, 2, 3, 4 (pre-lunch), 5.5, 8, 10 hours (pre-dinner) on Day 14
Population: The PK population was used which was defined as participants from the safety population who had plasma metformin, sitagliptin, and/or GSK2330672 PK parameter estimates from any portion of the study. Only those participants available at the specified time points were analyzed.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Groups:
- Sitagliptin 50 mg BID: Participants were randomized to receive solution of GSK2330672 90 mg orally BID for 14 days. Participants drank the contents of dosing bottle (45 mL) followed by 2×50 mL rinses of bottle and then an additional 95 mL water for a total volume of 240 mL consumed. The solution of GSK2330672 (2 mg/mL), was prepared by clinical staff pharmacists after reconstitution of GSK2330672 powder with phosphate buffer into amber glass bottles for administration. All dosing treatments, bottle rinses and additional water was consumed within a 15 minute period. Participants continued to receive metformin 850 mg tablet BID throughout the study (run-in and treatment period). Participants swallowed the whole metformin tablet with 240 mL of water and were instructed to avoid chewing or crushing.
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
Nanograms per milliliter (ng/mL) | 1102.2 (26.92) | 1289.3 (41.81) | 1219.9 (23.76) | 1160.0 (18.64) | 1378.8 (22.77) | 1376.6 (21.70) | 1223.5 (27.36)
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 10 mg BID; Test type: Superiority or Other — Each GSK2330672 dose level was compared to placebo using an analysis of variance (ANOVA) model of log-transformed values; Ratio = 1.17, 90% CI 2-sided [0.92 to 1.49] — Mean and confidence interval (CI) for the difference in least squares means (Active-Placebo) are back-transformed to form the point estimate and associated CI for the ratio of geometric means
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 20 mg BID; Test type: Superiority or Other — [test comment as in outcome 16, analysis 1]; Ratio = 1.11, 90% CI 2-sided [0.89 to 1.38] — Mean and CI for the difference in least squares means (Active-Placebo) are back-transformed to form the point estimate and associated CI for the ratio of geometric means
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 30 mg BID; Test type: Superiority or Other — [test comment as in outcome 16, analysis 1]; Ratio = 1.05, 90% CI 2-sided [0.87 to 1.27] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 60 mg BID; Test type: Superiority or Other — [test comment as in outcome 16, analysis 1]; Ratio = 1.25, 90% CI 2-sided [1.03 to 1.52] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Superiority or Other — [test comment as in outcome 16, analysis 1]; Ratio = 1.25, 90% CI 2-sided [1.04 to 1.50] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 50 mg BID; Test type: Superiority or Other — [test comment as in outcome 16, analysis 1]; Ratio = 1.11, 90% CI 2-sided [0.94 to 1.31] — [estimate comment as in outcome 16, analysis 2]

17. Secondary Outcome: PK Parameters for Metformin Steady State PK Parameters When Co-dosed With GSK2330672, Sitagliptin or Placebo-time of Occurrence of Cmax (Tmax)
Description: The time at which Cmax observed was determined directly from the raw concentration-time data.
Time Frame: as for outcome 16
Population: PK population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
Hour | 1.510 [1.00 to 4.00] | 1.000 [1.00 to 1.50] | 1.000 [0.50 to 3.98] | 1.050 [1.00 to 1.50] | 1.750 [0.50 to 4.00] | 1.500 [1.00 to 4.00] | 2.050 [1.00 to 4.02]

18. Secondary Outcome: PK Parameters for Metformin Steady State PK Parameters When Co-dosed With GSK2330672, Sitagliptin or Placebo-area Under the Concentration-time Curve Over the Dosing Interval of 10 Hours (AUC[0-10])
Description: PK population. Only those participants available at the specified time points were analyzed.
Time Frame: as for outcome 16
Population: PK population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour×ng/mL
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
Hour×ng/mL | 6805.8 (19.70) | 5982.0 (34.72) | 7066.2 (25.80) | 7066.5 (16.09) | 8090.5 (33.06) | 8375.3 (32.78) | 8425.4 (28.11)
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 10 mg BID; Test type: Superiority or Other — Each GSK2330672 dose level was compared to placebo using an ANOVA model following log-transformation; Ratio = 0.88, 90% CI 2-sided [0.68 to 1.13] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 20 mg BID; Test type: Superiority or Other — Each GSK2330672 dose level was compared to placebo using an ANOVA model following log-transformation; Ratio = 1.04, 90% CI 2-sided [0.82 to 1.31] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 30 mg BID; Test type: Superiority or Other — Each GSK2330672 dose level was compared to placebo using an ANOVA model following log-transformation; Ratio = 1.04, 90% CI 2-sided [0.85 to 1.26] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 60 mg BID; Test type: Superiority or Other — Each GSK2330672 dose level was compared to placebo using an ANOVA model following log-transformation; Ratio = 1.19, 90% CI 2-sided [0.97 to 1.45] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Superiority or Other — Each GSK2330672 dose level was compared to placebo using an ANOVA model following log-transformation; Ratio = 1.23, 90% CI 2-sided [1.01 to 1.49] — [estimate comment as in outcome 16, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 50 mg BID; Test type: Superiority or Other — Each GSK2330672 dose level was compared to placebo using an ANOVA model following log-transformation; Ratio = 1.24, 90% CI 2-sided [1.04 to 1.48] — [estimate comment as in outcome 16, analysis 2]

19. Secondary Outcome: Ratio to Baseline in Fasting Low-density Cholesterol (LDL) Cholesterol, High-density Cholesterol (HDL) Cholesterol, Total Cholesterol, Non-HDL Cholesterol and Triglycerides
Description: Data for fasting low-density cholesterol (LDL) cholesterol, high-density cholesterol (HDL) cholesterol, total cholesterol, non-HDL cholesterol and triglycerides is presented. Participants withdrawing early were excluded. Results were based on an ANCOVA model: Log(post-Baseline) - Log(Baseline) = Log(Baseline) + treatment + concomitant use of lipid lowering drugs.
Time Frame: Baseline (pre-dose Day -1) and Day 7, 14
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Ratio
  Cholesterol, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  Cholesterol, Day 7 | 0.95 (10.9) | 0.99 (12.1) | 0.84 (12.4) | 0.84 (13.7) | 0.74 (11.0) | 0.80 (3.7) | 0.97 (9.8)
  Cholesterol, Day 14: number analyzed (Participants) | 12 | 3 | 4 | 9 | 8 | 8 | 13
  Cholesterol, Day 14 | 0.95 (13.1) | 0.98 (14.2) | 0.81 (20.8) | 0.83 (18.5) | 0.75 (8.8) | 0.75 (6.7) | 0.92 (11.1)
  HDL cholesterol, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  HDL cholesterol, Day 7 | 1.00 (7.3) | 1.08 (12.8) | 1.05 (8.9) | 0.97 (8.0) | 0.95 (11.4) | 1.09 (15.7) | 0.97 (9.0)
  HDL cholesterol, Day 14: number analyzed (Participants) | 12 | 3 | 4 | 9 | 8 | 8 | 13
  HDL cholesterol, Day 14 | 0.99 (6.5) | 1.11 (1.5) | 1.02 (4.0) | 0.97 (8.8) | 0.96 (11.4) | 1.01 (11.6) | 0.97 (10.2)
  LDL cholesterol, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  LDL cholesterol, Day 7 | 0.97 (14.6) | 0.89 (6.4) | 0.77 (21.1) | 0.73 (21.5) | 0.58 (21.2) | 0.71 (6.5) | 1.00 (10.5)
  LDL cholesterol, Day 14: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  LDL cholesterol, Day 14 | 0.94 (17.6) | 0.80 (4.2) | 0.69 (23.1) | 0.72 (23.7) | 0.60 (15.0) | 0.67 (16.3) | 0.92 (15.3)
  Non-HDL Cholesterol, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  Non-HDL Cholesterol, Day 7 | 0.93 (13.8) | 0.96 (12.6) | 0.78 (18.2) | 0.80 (18.2) | 0.65 (12.0) | 0.73 (5.1) | 0.98 (11.9)
  Non-HDL Cholesterol, Day 14: number analyzed (Participants) | 12 | 3 | 4 | 9 | 8 | 8 | 13
  Non-HDL Cholesterol, Day 14 | 0.94 (17.7) | 0.94 (17.5) | 0.74 (29.7) | 0.78 (23.7) | 0.67 (7.2) | 0.68 (8.6) | 0.90 (15.1)
  Triglycerides, Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 8 | 9 | 13
  Triglycerides, Day 7 | 0.85 (20.6) | 1.07 (51.2) | 0.93 (18.8) | 1.11 (24.5) | 0.98 (19.8) | 0.93 (16.3) | 0.79 (32.7)
  Triglycerides, Day 14: number analyzed (Participants) | 12 | 3 | 4 | 9 | 8 | 8 | 13
  Triglycerides, Day 14 | 0.85 (23.0) | 1.21 (63.3) | 0.96 (35.8) | 1.07 (34.3) | 1.00 (16.6) | 1.00 (23.7) | 0.74 (34.5)
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — Results were based on an ANCOVA model: Log(post-Baseline) - Log(Baseline) = Log(Baseline) + treatment + concomitant use of lipid lowering drugs; Mean Difference (Net) = 1.03, 95% CI 2-sided [0.91 to 1.17] — Comparison for Day 7, cholesterol
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.88, 95% CI 2-sided [0.78 to 0.98] — Comparison for Day 7, cholesterol
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.86, 95% CI 2-sided [0.78 to 0.95] — Comparison for Day 7, cholesterol
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.75, 95% CI 2-sided [0.68 to 0.83] — Comparison for Day 7, cholesterol
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.83, 95% CI 2-sided [0.76 to 0.92] — Comparison for Day 7, cholesterol
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.01, 95% CI 2-sided [0.92 to 1.10] — Comparison for Day 7, cholesterol
Statistical Analysis 7: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.07, 95% CI 2-sided [0.95 to 1.19] — Comparison for Day 7, HDL cholesterol
Statistical Analysis 8: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.04, 95% CI 2-sided [0.94 to 1.16] — Comparison for Day 7, HDL cholesterol
Statistical Analysis 9: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.96, 95% CI 2-sided [0.88 to 1.05] — Comparison for Day 7, HDL cholesterol
Statistical Analysis 10: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.98, 95% CI 2-sided [0.89 to 1.07] — Comparison for Day 7, HDL cholesterol
Statistical Analysis 11: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.07, 95% CI 2-sided [0.98 to 1.17] — Comparison for Day 7, HDL cholesterol
Statistical Analysis 12: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.97, 95% CI 2-sided [0.90 to 1.05] — Comparison for Day 7, HDL cholesterol
Statistical Analysis 13: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.95, 95% CI 2-sided [0.80 to 1.13] — Comparison for Day 7, LDL cholesterol
Statistical Analysis 14: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.76, 95% CI 2-sided [0.65 to 0.90] — Comparison for Day 7, LDL cholesterol
Statistical Analysis 15: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.74, 95% CI 2-sided [0.64 to 0.85] — Comparison for Day 7, LDL cholesterol
Statistical Analysis 16: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.59, 95% CI 2-sided [0.51 to 0.69] — Comparison for Day 7, LDL cholesterol
Statistical Analysis 17: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.71, 95% CI 2-sided [0.62 to 0.81] — Comparison for Day 7, LDL cholesterol
Statistical Analysis 18: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.00, 95% CI 2-sided [0.89 to 1.14] — Comparison for Day 7, LDL cholesterol
Statistical Analysis 19: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.03, 95% CI 2-sided [0.88 to 1.21] — Comparison for Day 7, non-HDL cholesterol
Statistical Analysis 20: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.82, 95% CI 2-sided [0.71 to 0.95] — Comparison for Day 7, non-HDL cholesterol
Statistical Analysis 21: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.84, 95% CI 2-sided [0.74 to 0.95] — Comparison for Day 7, non-HDL cholesterol
Statistical Analysis 22: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.67, 95% CI 2-sided [0.59 to 0.76] — Comparison for Day 7, non-HDL cholesterol
Statistical Analysis 23: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.68 to 0.87] — Comparison for Day 7, non-HDL cholesterol
Statistical Analysis 24: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.02, 95% CI 2-sided [0.92 to 1.14] — Comparison for Day 7, non-HDL cholesterol
Statistical Analysis 25: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.27, 95% CI 2-sided [0.97 to 1.66] — Comparison for Day 7, triglycerides
Statistical Analysis 26: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.16, 95% CI 2-sided [0.90 to 1.50] — Comparison for Day 7, triglycerides
Statistical Analysis 27: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.30, 95% CI 2-sided [1.06 to 1.61] — Comparison for Day 7, triglycerides
Statistical Analysis 28: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.19, 95% CI 2-sided [0.96 to 1.48] — Comparison for Day 7, triglycerides
Statistical Analysis 29: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.15, 95% CI 2-sided [0.93 to 1.42] — Comparison for Day 7, triglycerides
Statistical Analysis 30: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.95, 95% CI 2-sided [0.79 to 1.16] — Comparison for Day 7, triglycerides
Statistical Analysis 31: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.00, 95% CI 2-sided [0.86 to 1.17] — Comparison for Day 14, cholesterol
Statistical Analysis 32: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.83, 95% CI 2-sided [0.73 to 0.96] — Comparison for Day 14, cholesterol
Statistical Analysis 33: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.82, 95% CI 2-sided [0.73 to 0.91] — Comparison for Day 14, cholesterol
Statistical Analysis 34: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.74, 95% CI 2-sided [0.66 to 0.82] — Comparison for Day 14, cholesterol
Statistical Analysis 35: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.69 to 0.86] — Comparison for Day 14, cholesterol
Statistical Analysis 36: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.93, 95% CI 2-sided [0.84 to 1.03] — Comparison for Day 14, cholesterol
Statistical Analysis 37: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.09, 95% CI 2-sided [0.99 to 1.21] — Comparison for Day 14, HDL cholesterol
Statistical Analysis 38: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.02, 95% CI 2-sided [0.93 to 1.11] — Comparison for Day 14, HDL cholesterol
Statistical Analysis 39: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.97, 95% CI 2-sided [0.90 to 1.04] — Comparison for Day 14, HDL cholesterol
Statistical Analysis 40: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.99, 95% CI 2-sided [0.92 to 1.06] — Comparison for Day 14, HDL cholesterol
Statistical Analysis 41: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.01, 95% CI 2-sided [0.94 to 1.08] — Comparison for Day 14, HDL cholesterol
Statistical Analysis 42: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.98, 95% CI 2-sided [0.92 to 1.04] — Comparison for Day 14, HDL cholesterol
Statistical Analysis 43: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.85, 95% CI 2-sided [0.69 to 1.04] — Comparison for Day 14, LDL cholesterol
Statistical Analysis 44: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.70, 95% CI 2-sided [0.58 to 0.85] — Comparison for Day 14, LDL cholesterol
Statistical Analysis 45: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.73, 95% CI 2-sided [0.62 to 0.86] — Comparison for Day 14, LDL cholesterol
Statistical Analysis 46: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.60, 95% CI 2-sided [0.50 to 0.71] — Comparison for Day 14, LDL cholesterol
Statistical Analysis 47: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.69, 95% CI 2-sided [0.59 to 0.80] — Comparison for Day 14, LDL cholesterol
Statistical Analysis 48: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.94, 95% CI 2-sided [0.81 to 1.09] — Comparison for Day 14, LDL cholesterol
Statistical Analysis 49: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.99, 95% CI 2-sided [0.80 to 1.22] — Comparison for Day 14, non-HDL cholesterol
Statistical Analysis 50: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.64 to 0.93] — Comparison for Day 14, non-HDL cholesterol
Statistical Analysis 51: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.67 to 0.90] — Comparison for Day 14, non-HDL cholesterol
Statistical Analysis 52: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.65, 95% CI 2-sided [0.55 to 0.75] — Comparison for Day 14, non-HDL cholesterol
Statistical Analysis 53: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.70, 95% CI 2-sided [0.60 to 0.81] — Comparison for Day 14, non-HDL cholesterol
Statistical Analysis 54: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.91, 95% CI 2-sided [0.80 to 1.04] — Comparison for Day 14, non-HDL cholesterol
Statistical Analysis 55: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.42, 95% CI 2-sided [1.01 to 2.00] — Comparison for Day 14, triglycerides
Statistical Analysis 56: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.28, 95% CI 2-sided [0.94 to 1.75] — Comparison for Day 14, triglycerides
Statistical Analysis 57: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.24, 95% CI 2-sided [0.98 to 1.58] — Comparison for Day 14, triglycerides
Statistical Analysis 58: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.22, 95% CI 2-sided [0.95 to 1.56] — Comparison for Day 14, triglycerides
Statistical Analysis 59: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 1.23, 95% CI 2-sided [0.96 to 1.57] — Comparison for Day 14, triglycerides
Statistical Analysis 60: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.89, 95% CI 2-sided [0.72 to 1.11] — Comparison for Day 14, triglycerides

20. Secondary Outcome: Ratio to Baseline in Fasting Apolipoprotein B
Description: Data for fasting apolipoprotein B is presented. Participants withdrawing early were excluded. Results were based on an ANCOVA model: Log(post-Baseline) - Log(Baseline) = Log(Baseline) + treatment + concomitant use of lipid lowering drugs.
Time Frame: Baseline (pre-dose Day -1) and Day 7, 14
Population: Safety population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13 | 5 | 5 | 9 | 9 | 10 | 13
Ratio
  Day 7: number analyzed (Participants) | 12 | 4 | 5 | 9 | 7 | 9 | 13
  Day 7 | 0.97 (10.6) | 0.95 (5.9) | 0.78 (13.9) | 0.81 (13.1) | 0.69 (12.0) | 0.76 (3.8) | 0.96 (10.3)
  Day 14: number analyzed (Participants) | 12 | 4 | 4 | 9 | 7 | 8 | 13
  Day 14 | 0.93 (14.2) | 0.85 (6.7) | 0.75 (19.0) | 0.78 (19.6) | 0.67 (14.9) | 0.69 (9.3) | 0.88 (15.5)
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.98, 95% CI 2-sided [0.87 to 1.11] — Comparison for Day 7, apolipoprotein B
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.79, 95% CI 2-sided [0.71 to 0.89] — Comparison for Day 7, apolipoprotein B
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.82, 95% CI 2-sided [0.74 to 0.90] — Comparison for Day 7, apolipoprotein B
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.70, 95% CI 2-sided [0.63 to 0.77] — Comparison for Day 7, apolipoprotein B
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.70 to 0.85] — Comparison for Day 7, apolipoprotein B
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.97, 95% CI 2-sided [0.89 to 1.06] — Comparison for Day 7, apolipoprotein B
Statistical Analysis 7: Comparison: Placebo vs GSK2330672 10 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.91, 95% CI 2-sided [0.77 to 1.07] — Comparison for Day 14, apolipoprotein B
Statistical Analysis 8: Comparison: Placebo vs GSK2330672 20 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.81, 95% CI 2-sided [0.68 to 0.95] — Comparison for Day 14, apolipoprotein B
Statistical Analysis 9: Comparison: Placebo vs GSK2330672 30 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.80, 95% CI 2-sided [0.70 to 0.91] — Comparison for Day 14, apolipoprotein B
Statistical Analysis 10: Comparison: Placebo vs GSK2330672 60 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.67, 95% CI 2-sided [0.58 to 0.77] — Comparison for Day 14, apolipoprotein B
Statistical Analysis 11: Comparison: Placebo vs GSK2330672 90 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.73, 95% CI 2-sided [0.64 to 0.83] — Comparison for Day 14, apolipoprotein B
Statistical Analysis 12: Comparison: Placebo vs Sitagliptin 50 mg BID; An estimation approach was used; Test type: Superiority or Other — [test comment as in outcome 19, analysis 1]; Mean Difference (Net) = 0.90, 95% CI 2-sided [0.80 to 1.02] — Comparison for Day 14, apolipoprotein B

21. Secondary Outcome: Sitagliptin Steady State PK Parameters When Co-dosed With Metformin-Cmax Following the First and Second Sitagliptin Doses
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data following the first and second dose of sitagliptin on Day 14 (Cmax1 and Cmax2).
Time Frame: Fasting pre-dose (within 15 minutes of dose), 1, 2, 3, 4 (pre-lunch), 10 (pre-dinner), 13 and 14 hours (bed time) on Day 14
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ng/mL
Arm/Group | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13
Ng/mL
  Cmax 1 | 238.2 (26.20)
  Cmax 2 | 188.5 (25.34)

22. Secondary Outcome: Sitagliptin Steady State PK Parameters When Co-dosed With Metformin-Tmax Following the First and Second Sitagliptin Doses
Description: The time at which Cmax was observed by determining directly from the raw concentration-time data following the first and second dose of sitagliptin on Day 14 (Tmax1 and Tmax2). If data permits, Tmax2 was defined as the time of Cmax following the second dose of sitagliptin.
Time Frame: as for outcome 21
Population: PK population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13
Hour
  Tmax 1 | 2.000 [1.00 to 3.98]
  Tmax 2 | 3.050 [2.98 to 4.07]

23. Secondary Outcome: Sitagliptin Steady State PK Parameters When Co-dosed With Metformin-AUC(0-10)
Description: The AUC(0-10) following the first dose and prior to the second dose of sitagliptin was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Fasting pre-dose (within 15 minutes of dose), 1, 2, 3, 4 (pre-lunch), 10 (pre-dinner) on Day 14
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour×ng/mL
Arm/Group | Sitagliptin 50 mg BID
Number analyzed (Participants) | 13
Hour×ng/mL | 1473.5 (22.45)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from run-in period until the follow-up contact (7-10 days after discharge). SAEs and non-SAE were reported from treatment period only (up to 14 days).
Description: Safety population used for assessment of safety results.
Arm/Group | Placebo | GSK2330672 10 mg BID | GSK2330672 20 mg BID | GSK2330672 30 mg BID | GSK2330672 60 mg BID | GSK2330672 90 mg BID | Sitagliptin 50 mg BID
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/5 | 0/5 | 0/9 | 0/9 | 0/10 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/5 | 0/5 | 0/9 | 0/9 | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 9/13 | 3/5 | 5/5 | 5/9 | 8/9 | 8/10 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | GSK2330672 10 mg BID (N=5) | GSK2330672 20 mg BID (N=5) | GSK2330672 30 mg BID (N=9) | GSK2330672 60 mg BID (N=9) | GSK2330672 90 mg BID (N=10) | Sitagliptin 50 mg BID (N=13)
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | GSK2330672 10 mg BID (N=5) | GSK2330672 20 mg BID (N=5) | GSK2330672 30 mg BID (N=9) | GSK2330672 60 mg BID (N=9) | GSK2330672 90 mg BID (N=10) | Sitagliptin 50 mg BID (N=13)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 5 | 2 | 7 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 1 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 3 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scleral hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.